CLINICAL TRIAL: NCT00275951
Title: Phase II Study of Cetuximab Plus P-HDFL(Cisplatin and Weekly 24-Hour Infusion of High-dose 5-Fluorouracil and Leucovorin)for the First-line Treatment of Advanced Gastric Cancer
Brief Title: Cetuximab Plus P-HDFL for the First-line Treatment of Advanced Gastric Cancer
Acronym: FLAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other); Chang Gung Memorial Hospital (Other); Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 941004
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Gastric Cancer
Keywords: Combination; Chemotherapy; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab Plus P-HDFL (Experimental): Cetuximab 400 mg/m2, IV, day 1 of cycle 1; then weekly IV 250 mg/m2. Cisplatin 24-hour IV infusion 35 mg/m2/day, plus HDFL (5-FU 2,000 mg/m2 and leucovorin 300 mg/m2), day 1 and day 8. HDFL IV, day 15.
  Interventions: Drug: Cetuximab Plus P-HDFL

INTERVENTIONS:
Drug: Cetuximab Plus P-HDFL — Cetuximab 400 mg/m2, IV, day 1 of cycle 1; then weekly IV 250 mg/m2. Cisplatin 24-hour IV infusion 35 mg/m2/day, plus HDFL (5-FU 2,000 mg/m2 and leucovorin 300 mg/m2), day 1 and day 8. HDFL IV, day 15.

SUMMARY:
The investigators have initial evidence that the combination of cetuximab and cisplatin-HDFL may further improve the efficacy of the cisplatin-HDFL combination chemotherapy.

DETAILED DESCRIPTION:
The clinical efficacy (confirmed objective response rates, progression-free survival, overall survival), and treatment-related toxicities of this novel regimen will be examined as the first-line treatment in patients with nonresectable or recurrent/metastatic gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years
2. Histologically proven adenocarcinoma
3. At least one "measurable" lesion (by RECIST)
4. No prior chemotherapy for gastric cancer
5. WHO performance status ≦ 2
6. Adequate baseline organ functions
7. Fasting serum triglyceride level > 70 mg/dL
8. Written informed consent
9. At least one month from gastrectomy
10. Availability of tumor sample for immunohistochemical or pharmacogenomic testing of EGFR

Exclusion Criteria:

1. Concomitant anti-cancer biological agents, chemotherapy, or radiotherapy
2. CNS metastasis
3. Pregnancy, breast-feeding women and women of child-bearing potential
4. Life expectancy less 3 months
5. Serious concomitant illness
6. Concurrent or prior second malignancy
7. Known hypersensitivity reaction to any of the components of study treatments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Confirmed objective response rates | Confirmed objective response within 4 weeks

SECONDARY OUTCOMES:
Progression-free survival (PFS), overall survival (OS), treatment-related toxicity | 3 years and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Lii Cheng, M.D., Ph.D., Study Chair — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan